CLINICAL TRIAL: NCT05865691
Title: Role of Coagulation, Inflammation and Vessels in Chronic Liver Disease
Acronym: CLUE
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220750; 2022-A01421-42 (Other: IDRCB)
Record Dates: First submitted 2023-04-24; First posted 2023-05-19 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Chronic Liver Diseases; Coagulation
MeSH Terms: conditions — Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- controls without liver disease: blood collection on the day of inclusion
  Interventions: Other: biomarker assay
- patients with chronic liver disease without cirrhosis: blood collection on the day of inclusion
  Interventions: Other: biomarker assay
- patients with chronic liver disease with compensated cirrhosis: blood collection on the day of inclusion
  Interventions: Other: biomarker assay
- patients with chronic liver disease with stable decompensated cirrhosis: blood collection on the day of inclusion
  Interventions: Other: biomarker assay
- patients with chronic liver disease with decompensated cirrhosis in the acute phase: blood collection on the day of inclusion
  Interventions: Other: biomarker assay
- patients with chronic liver disease with decompensated cirrhosis and organ failure: blood collection on the day of inclusion
  Interventions: Other: biomarker assay

INTERVENTIONS:
Other: biomarker assay — blood sample on the day of inclusion
  Other Names: blood sample

SUMMARY:
Chronic liver diseases represent a major public health problem and are responsible for more than 150,000 deaths in Europe each year. These diseases are accompanied by symptoms that profoundly alter the quality of life and mainly affect people of working age, leading to a major economic impact.

Coagulation disorders, inflammation and vascular alterations are associated with chronic liver diseases but their role in the onset and/or progression of liver diseases is still not fully understood.

A better understanding of chronic liver diseases and in particular of the factors that play a role in the onset and progression of these diseases would improve patient management and therefore have a positive impact on individuals, but also on the healthcare system and the economy.

DETAILED DESCRIPTION:
Chronic liver diseases represent a major public health problem and are responsible for more than 150,000 deaths in Europe each year. These diseases are accompanied by symptoms that profoundly alter the quality of life and mainly affect people of working age, leading to a major economic impact.

Coagulation disorders, inflammation and vascular alterations are associated with chronic liver diseases but their role in the onset and/or progression of liver diseases is still not fully understood.

A better understanding of chronic liver diseases and in particular of the factors that play a role in the onset and progression of these diseases would improve patient management and therefore have a positive impact on individuals, but also on the healthcare system and the economy.

The main objective is to identify the role of coagulation in the development and progression of chronic liver diseases and their complications.

ELIGIBILITY:
Inclusion Criteria:

Patients with chronic liver disease:

Patients over 18 years of age Patients affiliated with a social security plan or entitled to receive benefits Patients with chronic liver disease or cirrhosis whose diagnosis is based on one or more of the following

* Liver biopsy showing chronic liver disease or cirrhosis
* Liver elastography by Fibroscan® assessing the elasticity of the liver at more than 10 kpa
* Combination of clinical, biological and imaging criteria characteristic of chronic liver disease (signs of portal hypertension, liver failure and liver dysmorphia in a patient with at least one risk factor for chronic liver disease)

Controls without liver disease Patients 18 years of age with no known liver disease Patients who have had blood drawn in the hospital prior to surgery (pre-operative work-up as part of the care process).

Exclusion Criteria:

Common non-inclusion criteria for patients with chronic liver disease and controls without liver disease will be as follows:

* Pregnant or lactating women
* Protected populations: persons under guardianship, under curatorship or safeguard of justice
* Patient under AME
* Patient who has not signed a consent form
* Recent surgery before the blood test (< 2 weeks)
* Transfusion of blood products (packed red blood cells, platelet concentrates, fresh frozen plasma, etc.) recently (< 2 weeks)
* Use of medication that interferes with hemostasis
* Active extra-hepatic cancer or cancer less than 5 years old
* Organ transplantation (liver, kidney, lung, heart)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age with chronic liver disease Controls without liver disease will be individuals over 18 years of age without liver disease
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2035-10-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Activated partial thromboplastin time abnormalities in patients with chronic liver disease at different stages and controls without liver disease | at 10 years
  Mesure of activated partial thromboplastin time for each patient at inclusion
Factor II abnormalities in patients with chronic liver disease at different stages and controls without liver disease | at 10 years
  Mesure of factor II for each patient at inclusion
Factor V abnormalities in patients with chronic liver disease at different stages and controls without liver disease | at 10 years
  Mesure of factor V for each patient at inclusion
Factor VII abnormalities in patients with chronic liver disease at different stages and controls without liver disease | at 10 years
  Mesure of factor VII for each patient at inclusion
Factor VIII abnormalities in patients with chronic liver disease at different stages and controls without liver disease | at 10 years
  Mesure of factor VIII for each patient at inclusion
Factor IX abnormalities in patients with chronic liver disease at different stages and controls without liver disease | at 10 years
  Mesure of factor IX for each patient at inclusion
Factor X abnormalities in patients with chronic liver disease at different stages and controls without liver disease | at 10 years
  Mesure of factor X for each patient at inclusion
Factor XI abnormalities in patients with chronic liver disease at different stages and controls without liver disease | at 10 years
  Mesure of factor XI for each patient at inclusion
Fibrinogen abnormalities in patients with chronic liver disease at different stages and controls without liver disease | at 10 years
  Mesure of fibrinogen for each patient at inclusion
D-dimer abnormalities in patients with chronic liver disease at different stages and controls without liver disease | at 10 years
  mesure of D-dimer for each patient at inclusion
Protein C abnormalities in patients with chronic liver disease at different stages and controls without liver disease | at 10 years
  Mesure of protein C for each patient at inclusion
protein S abnormalities in patients with chronic liver disease at different stages and controls without liver disease | at 10 years
  mesure of protein S for each patient at inclusion
Willebrand factor abnormalities in patients with chronic liver disease at different stages and controls without liver disease | at 10 years
  Mesure of plasma Willebrand factor for each patient at inclusion
Thrombin generation test abnormalities in patients with chronic liver disease at different stages and controls without liver disease | at 10 years
  Mesure of thrombin generation test for each patient at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Emmanuel Rautou, Principal Investigator — APHP
Locations (1):
- Beaujon Hospital, Clichy, France